CLINICAL TRIAL: NCT03314896
Title: Laparoscopic Surgery for T4 Tumor of the Colon Cancer: A Prospective, MultiCenter, Randomized, Open-Label, Parallel Group Clinical Trial (LST4C Trial)
Brief Title: Laparoscopic Surgery for T4 Tumor of the Colon Cancer (LST4C Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LI XIN-XIANG (Other)
Responsible Party: Sponsor-Investigator, LI XIN-XIANG, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LST4C trial
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Colonic Neoplasms
Keywords: Colonic Neoplasms; Laparoscopic Surgery; T4
MeSH Terms: conditions — Colonic Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic surgery for T4 colon tumor (Experimental): Laparoscopic surgery for T4 colon cancers
  Interventions: Procedure: Laparoscopic surgery
- Open surgery for T4 colon tumor (No Intervention): Conventional open surgery for T4 colon cancers

INTERVENTIONS:
Procedure: Laparoscopic surgery
  Other Names: Laparoscopic surgery for T4 colon cancers
  Arms: Laparoscopic surgery for T4 colon tumor

SUMMARY:
The purpose of this study is to compare the short- and long-term survival of laparoscopic surgery and conventional open surgery for T4 colon cancer

DETAILED DESCRIPTION:
The investigators previous study indicated that laparoscopic surgery is feasible in T4 colon cancers with comparable clinical and oncologic outcomes. Laparoscopy can be considered as an alternative approach for T4 colon cancers with the advantage of faster recovery. However, the clinical value of laparoscopic surgery for T4 colon cancer was only validated in some retrospective study and some prospective study in single institute with small sample of patients. The aim of the present study is to compare the short-and long-term survival outcomes of laparoscopic surgery and conventional open surgery for T4 colon cancer as well as the mortality and the morbidity. The number of patients needed to get a 80% power is 1960. The average number of patients/surgical center is approximately 200 in each of 10 surgical centers. The preoperative, intraoperative and postoperative period will be in complete accordance with the usual care of the center. The baseline demographics and conditions as well as the perioperative items and the postoperative occurrences will be recorded through a prior designed equestionnaire.

Systematically analyze and compare the disease free survival rate, the mortality, the morbidity, and the proportion of completion of laparoscopic surgery of the two surgical strategies (laparoscopy VS conventional open surgery).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent

  * Histologically confirmed diagnosis of colon carcinoma
  * CT or MRI verified as T4 colon cancer without involvement of other organs
  * Without multiple lesion other than carcinoma in situ
  * Tumor size < 8 cm
  * No bowel obstruction
  * Sufficient organ function
  * No history of gastrointestinal surgery
  * 18 years of age or older
  * Performance Status (ECOG) 0, 1 or 2 and life expectancy > 12 weeks
  * Operable patients

Exclusion Criteria:

* • Women who are pregnant (confirmed by serum b-HCG in women of reproductive age) or breast feeding

  * Unstable or uncompensated respiratory or cardiac disease
  * Serious active infections
  * Hypersensitivity to capecitabine/fluorouracil or oxaliplatin
  * Stomatitis, ulceration in the mouth or gastrointestinal tract
  * Severe diarrhea
  * Peripheral sensory neuropathy with functional impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 957 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3-year
  calculated from the date of diagnosis to the date of death from any cause

SECONDARY OUTCOMES:
Disease free survival | 3-year
  calculated from the date of surgery to the date of recurrence
Adverse events (mortality and morbidity) | 3-month
  Number of participants with treatment-related adverse events assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Xinxiang Li, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No